CLINICAL TRIAL: NCT06754410
Title: Efficacy of Antihistamine Drugs as Medical Expulsive Therapy Alone or in Combination With Alpha Blockers: A Prospective Randomized Controlled Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mostafa AbdelRazek, Assistant Professor of Urology, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SVU.MED.URO016.4.23,5,638
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Lower Ureteric Stones
Keywords: stones , ureter, tamsulosin
MeSH Terms: conditions — Calculi | interventions — Tamsulosin; Cetirizine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tamsulosin (Active Comparator): All patients of group A received tamsulosin 0.4 mg once daily
  Interventions: Drug: Tamsulosin
- Cetirizine (Active Comparator): All patients of group B received Cetirizine once daily
  Interventions: Drug: Cetirizine
- Cetirizine + Tamsulosin (Active Comparator): All patients of group C received Tamsulosin 0.4 mg and Cetirizine once daily
  Interventions: Combination Product: Cetirizine + Tamsulosin
- Placebo (Placebo Comparator): All patients of group D received Placebo once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tamsulosin — group A take tamsulosin once daily
  Arms: Tamsulosin
Drug: Cetirizine — give cetirizine once dailly
  Arms: Cetirizine
Combination Product: Cetirizine + Tamsulosin — both once daily
  Arms: Cetirizine + Tamsulosin
Other: Placebo — once dailly
  Arms: Placebo

SUMMARY:
we investigate the Efficacy of Antihistamine Drugs as Medical Expulsive Therapy Alone or in Combination with Alpha Blockers in distal ureter stone

ELIGIBILITY:
Inclusion Criteria:

* all adult patients with lower ureter stone less than 10 mm

Exclusion Criteria:

* pregnant, solitary kidney, sensitivity to drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
ureter stone free rate | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Qena university hospital, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR